CLINICAL TRIAL: NCT07146815
Title: PolyCystic Ovary Syndrome as Suggested Risk Group for Non-Alcoholic Fatty Liver Disease
Acronym: P-CORIGA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Z-2022027
Record Dates: First submitted 2025-07-29; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-07

CONDITIONS: NAFLD (Nonalcoholic Fatty Liver Disease); Polycystic Ovarian Syndrome (PCOS)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCOS group (Other): Screening of women with PCOS
  Interventions: Diagnostic Test: FibroScan; Diagnostic Test: MRI PDFF
- Control group (Other): Screening of women without PCOS
  Interventions: Diagnostic Test: FibroScan; Diagnostic Test: MRI PDFF

INTERVENTIONS:
Diagnostic Test: FibroScan — Performance of a FibroScan measurement to determine the prevalence of liver steatosis.
Diagnostic Test: MRI PDFF — Performance of an MRI-PDFF to determine amount of liver steatosis.

SUMMARY:
To study the prevalence, non-invasive diagnostics and evolution of non-alcoholic-fatty-liver-disease (NAFLD) in patients with polycystic ovary syndrome (PCOS)

ELIGIBILITY:
Inclusion Criteria:

* Adults (i.e. older than 18 years of age)
* The diagnosis of PCOS based on expert opinion (i.e. according to Rotterdam criteria)
* Able to understand patients information concerning this study
* Able to give written informed consent

Exclusion Criteria:

* Excessive alcohol use: ≥ 2u (20g)/day for females
* Exclusion of other causes of liver disease
* Secondary causes of liver steatosis
* Other causes of endocrinological disease
* Diseases that might mimic PCOS

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 157 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of NAFLD | Baseline and at follow-up 1 year later.
  To study the prevalence of NAFLD in a population diagnosed with PCOS measured with Controlled Attenuation Parameter (CAP)
Prevalence of NAFLD in PCOS | Baseline
  To measure the prevalence of NAFLD in women with PCOS using the MRI-PDFF technique.

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: Undecided